CLINICAL TRIAL: NCT00157300
Title: PROTECT: Prospective Trial on Erythropoietin in Clinical Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Ton Rabelink, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P05-026
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Patients Receiving a Kidney From a Non-Heart-Beating Donor
Keywords: erythropoietin; kidney transplantation; delayed graft function
MeSH Terms: conditions — Delayed Graft Function | interventions — epoetin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epoetin beta (Experimental)
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — intravenous, 33000 IU, 3 consecutive days, starting 3-4 hours before transplantation. Total dose 100.000 IU.
  Other Names: Neorecormon

SUMMARY:
Randomized, double blind, placebo controlled, prospective trial investigating the effect of erythropoietin in renal transplantation.

The investigators postulate that erythropoietin reduces the risk of delayed graft function.

DETAILED DESCRIPTION:
Randomized, double blind, placebo controlled, prospective trial in patients, receiving a kidney transplantation. Patients will be randomized to receive either Epoetin Beta (Neorecormon; Roche) or placebo.

The primary endpoint will be delayed graft function. The anticipated duration of this trial is 2 year and the target sample size is 60 patients per arm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Receiving a kidney from a non-heart-beating donor category 3

Exclusion Criteria:

* Donor related factors: a prolonged warm ischaemic time (> 45 min); a cold ischaemic time of > 24 hours; serum creatinin of > 150 umol/l

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-07; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
incidence of delayed graft function and primary non function after kidney transplantation | within12 weeks after transplantation

SECONDARY OUTCOMES:
duration of dialysis treatment | within 12 weeks after transplantation
incidence of acute rejection episodes | till one year after transplantation
renal function at 3, 6 and 12 months | 3, 6 and 12 months after transplantation
patient and graft survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ton Rabelink, MD, PhD, Study Chair — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Other transplantation centers, To Be Determined

REFERENCES:
- [Background] Ehrenreich H, Hasselblatt M, Dembowski C, Cepek L, Lewczuk P, Stiefel M, Rustenbeck HH, Breiter N, Jacob S, Knerlich F, Bohn M, Poser W, Ruther E, Kochen M, Gefeller O, Gleiter C, Wessel TC, De Ryck M, Itri L, Prange H, Cerami A, Brines M, Siren AL. Erythropoietin therapy for acute stroke is both safe and beneficial. Mol Med. 2002 Aug;8(8):495-505. PMID 12435860
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280